CLINICAL TRIAL: NCT03248401
Title: Effect of Cilostazol, a Phosphodiesterase 3 Inhibitor, on Carotid Atherosclerosis Estimated by 3D Ultrasound in Patients With Type 2 Diabetes
Brief Title: Effect of Cilostazol on Carotid Atherosclerosis Estimated by 3D Ultrasound in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Soo Lim, Professor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Cilostazol_Carotid a. plaque
Record Dates: First submitted 2017-08-09; First posted 2017-08-14 (Actual); Last update posted 2020-04-08 (Actual); Status verified 2020-04

CONDITIONS: Type 2 Diabetes Mellitus; Carotid Atherosclerosis
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Carotid Artery Diseases | interventions — Cilostazol; Aspirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cilostazol group (Experimental): Cilostazol 200 mg or maximal tolerate dose
  Interventions: Drug: Cilostazol
- Aspirin group (Active Comparator): Aspirin 100 mg
  Interventions: Drug: Aspirin

INTERVENTIONS:
Drug: Cilostazol — Cilostazol 200 mg/day
  Arms: Cilostazol group
Drug: Aspirin — Aspirin 100 mg/day
  Arms: Aspirin group

SUMMARY:
To investigate the effect of cilostazol compared with aspirin on carotid atherosclerosis in patients with type 2 diabetes mellitus

ELIGIBILITY:
Inclusion Criteria:

* Age between 30 and 80 years
* Patients with type 2 diabetes on treatment (HbA1c 6.0-11.0%)
* Carotid plaque on 3D ultrasound

Exclusion Criteria:

* Acute bleeding or bleeding tendency
* Diagnosed with heart failure
* Suggestive of ischemia on ECG
* Uncontrolled hypertension
* Recently diagnosed with peptic ulcer disease
* Taking other antiplatelet agents
* Hypersensitivity to salicylic acid
* Aspirin induced asthma
* Severe kidney, liver, heart disease

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-09-26 (Actual); Primary Completion 2018-10-21 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Change of carotid artery atherosclerosis | 6 months
  Plaque composition

SECONDARY OUTCOMES:
Change of carotid artery atherosclerosis 1 | 6 months
  Changes in carotid intima-media thickness after treatment
Change of carotid artery atherosclerosis 2 | 6 months
  Changes in carotid artery stenosis after treatment
Change of carotid artery atherosclerosis 3 | 6 months
  Plaque volume in carotid artery

OTHER OUTCOMES:
Glucose metabolism 1 | 6 months
  HOMA-Insulin Resistance
Diabetic complication | 6 months
  Albuminuria
Glucose metabolism 2 | 6 months
  HbA1c
Body composition | 6 months
  Body fat mass and percent

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

REFERENCES:
- [Background] Katakami N, Kim YS, Kawamori R, Yamasaki Y. The phosphodiesterase inhibitor cilostazol induces regression of carotid atherosclerosis in subjects with type 2 diabetes mellitus: principal results of the Diabetic Atherosclerosis Prevention by Cilostazol (DAPC) study: a randomized trial. Circulation. 2010 Jun 15;121(23):2584-91. doi: 10.1161/CIRCULATIONAHA.109.892414. Epub 2010 Jun 1. PMID 20516379
- [Background] Huh JH, Seok H, Lee BW, Kang ES, Lee HC, Cha BS. Effect of cilostazol on carotid intima-media thickness in type 2 diabetic patients without cardiovascular event. Endocrine. 2014 Sep;47(1):138-45. doi: 10.1007/s12020-013-0120-y. Epub 2014 Jan 1. PMID 24381128
- [Derived] Lee DH, Chun EJ, Moon JH, Yun HM, Lim S. Effect of cilostazol on carotid plaque volume measured by three-dimensional ultrasonography in patients with type 2 diabetes: The FANCY study. Diabetes Obes Metab. 2020 Dec;22(12):2257-2266. doi: 10.1111/dom.14147. Epub 2020 Sep 17. PMID 32700396